CLINICAL TRIAL: NCT03139994
Title: One Habitual Chewing Side May Contribute to Chronic Temporomandibular Joint Disorder Pain
Brief Title: Altered MAstication Contribute to TMJ PAin
Acronym: MAPA
Status: Completed | Type: Observational
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Urbano Santana Penin, MD, DDS, PhD, PROFESSOR, University of Santiago de Compostela
Other Study IDs: 20130123
Record Dates: First submitted 2016-05-10; First posted 2017-05-04 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Temporomandibular Joint Disorders; Mastication Disorder
Keywords: occlusion; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bites and Stings; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Diagnostic — OBSERVATIONAL, DIAGNOSTIC PROCEDURES. Young adults with no signs or symptoms of TMD will be assessed. The chewing function, condylar path angles and lateral guidance angles will be recorded. Maximum comfortable and unassisted jaw opening, hemispheric dominance and hemimandibular retrognathia will be considered as secondary pre-specified outcomes. Three-Four years later, both TMJs of each participant presenting signs and/or symptoms will be evaluated according to DC/TMD. Same recordings as baseline will be carried out.

SUMMARY:
The cause of temporomandibular joint disorders remains unknown. It is considered multifactorial and includes physical (peripheral) and psychosocial (central) factors. It has been showed an association: a steeper condylar path, flatter lateral anterior guidance, and habitual chewing on the symptomatic side. This finding argues the possibility of causation of some of these characteristics. This double blind longitudinal study aims to assess if the presence of one habitual chewing side could contribute to temporomandibular joint disorders over time.

Method. Young adults with no signs or symptoms of TMD will be assessed. Participants with one chewing side (observed and interview); with steeper condylar path and lower lateral guidance angles will be considered consistent one side chewers, and this side will be considered more susceptible to suffer TMD. Mouth opening, hemispheric dominance and hemimandibular retrognathia will be considered as secondary pre-specified outcomes. Four years later, both TMJs of each participant presenting signs and/or symptoms will be evaluated according to DC/TMD.

ELIGIBILITY:
Inclusion Criteria:

* healthies
* full dentates
* normal occlusion
* One habitual chewing side

Exclusion Criteria:

* Severe malocclusion, dental decay, severe periodontal disease.

Pains from other origins or Orthodontics are not criteria for exclusion

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical or Dental School students. Healthy young adults with fully dentate normal occlusion
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Presence or not of symptoms of temporomandibular joint disorders according to DC/TMD | At 3 years follow-up
  Pain-intensity (0-10 VAS scale, Von Korf)
Change of maximal unassited jaw opening | Baseline and 3 years follow-up
  Maximum unassisted jaw opening or interincisal distance (from edge to edge) measured by a Boley gauge. Up 38 in females and up 40 mm in males are considered limited.

SECONDARY OUTCOMES:
Change of condylar paths angles inclination | Baseline and 3-4-years follow-up (end of the study)
  Alteration of parasagittal plane Axiography of condyle motion in respect Frankfort horizontal plane
Alteration of lateral dental guidance angles | Baseline and 4-years follow-up (end of the study)
  Angle between Frankfort plane and lateral dental anterior guidance
Change of maximal comfortable jaw opening | Baseline and 4-years follow-up (end of the study)
  Maximum jaw opening or interincisal distance (from edge to edge) measured by a Boley gauge. Up 38 in females and up 40 mm in males are considered limited.
Change of the habitual chewing side | Baseline and 3-4-years follow-up (end of the study)
  Determining the habitual chewing side by direct observation using chewing gum, First cicle, and subsequent cicles (7 or over of 10 cicles), interview (used one habitual chewing side?: 1, no, alternate; 2, yes, right; 3, yes, left; 4, I don't know) and kinesiography.
Change of lateral deviation during maximal unassisted jaw opening | Baseline, 3 years follow-up
  Kiesiography K7

OTHER OUTCOMES:
Hemimandibular retrognathia | Baseline
  Interincisal median midline and Angle Class on each side
Hemispheric dominance, asuming oposite side to handedness preference | Baseline
  Edinburg inventory (Oldfield)
Change of Life quality | Baseline, 3 years follow-up
  SCL-90-R self-administered questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Urbano Santana-Mora, PhD, Principal Investigator — University of Santiago de Compostela. Spain; Urbano Santana, Prof., Study Chair — University of Santiago de Compostela. Spain; Mª Jesús Mora, Principal Investigator — University of Santiago de Compostela. Spain
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in a on-line appendix linked from the article in a JCR Journal.

REFERENCES:
- [Result] Santana-Mora U, Lopez-Cedrun J, Mora MJ, Otero XL, Santana-Penin U. Temporomandibular disorders: the habitual chewing side syndrome. PLoS One. 2013 Apr 8;8(4):e59980. doi: 10.1371/journal.pone.0059980. Print 2013. PMID 23593156